CLINICAL TRIAL: NCT07117409
Title: Retrospective Observational Study on the Safety of Nivolumab in Patients With Metastatic Renal Carcinoma and Renal Failure
Brief Title: Retrospective Study on the Safety of Nivolumab in Patients With mRCC and Renal Failure
Acronym: RI-NIVO
Status: Terminated | Type: Observational
Why Stopped: Healted Prematurely
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 622/2019/OSS/IRCCSRE
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: renal failure; carcinoma; nivolumab
MeSH Terms: conditions — Carcinoma, Renal Cell; Renal Insufficiency; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with normal or mildly reduced renal function (GFR<90 and ≥60 ml/min/1.73 m^2)
- Patients with moderate renal failure (GFR <60 e ≥30 ml/min/1.73 m^2)
- Patients with severe renal failure (GFR <30 e ≥15 ml/min/1.73 m^2)

SUMMARY:
This is an observational, retrospective, multicenter study aimed to compare the toxicity of Nivolumab in patients with metastatic renal cell carcinoma treated in line II and III stratified into 3 patient groups:

* patients with normal or mildly reduced renal function (GFR<90 and ≥60 ml/min/1.73 m^2);
* patients with moderate renal impairment (GFR <60 e ≥30 ml/min/1.73 m^2),
* patients with severe renal impairment (GFR <30 e ≥15 ml/min/1.73 m^2) Patients must have been treated with Nivolumab, as per clinical practice. All patients who have received at least one drug administration between february 2017 to December 31, 2018 will be enrolled in the study.

DETAILED DESCRIPTION:
The treatment of metastatic renal cancer has undergone several changes in recent years especially regarding second line treatment which has seen the development of new ones antiangiogenic drugs such as cabozantinib and immunotherapy with inhibitory checkpoints (nivolumab). Nivolumab is a human IgG4 monoclonal antibody that binds to the receptor 'programmed-death' 1 (PD-1) by blocking its interaction with its ligand (PD-L1). The PD-1 receptor has an action negative regulatory on T lymphocyte activity, the interaction between receptor and ligand (PD-L1) expressed by cancer cells involves inhibition of T cell proliferation and cytokine secretion. The metabolism of Nivolumab was not well characterized, although it is probably degraded into small peptides and amino acids through catabolic pathways similar way to endogenous IgG; all this is important as there is no involvement by normal excretory/emuntory organs such as liver and kidney. The patient affected by metastatic renal cell carcinoma presents more frequently than a subject of the same sex and age a picture of concomitant renal insufficiency (IR); this data could be linked to age median at diagnosis (65 years), high incidence of diabetes and arterial hypertension, and presence of a previous nephrectomy .Renal impairment (IR) is classified as: - mild (glomerular filtrate (GFR) <90 and ≥60 ml/min/1.73 m^2); - moderate (GFR <60 and ≥30 ml/min/1.73 m^2), or severe (GFR <30 and ≥15 ml/min/1.73 m^2) Some pharmacokinetic analyses have been conducted for patients with mild renal impairment or moderate who have not documented clinically detected differences in clearance of Nivolumab compared to patients with normal renal function; however this is a number very modest number of patients with moderate IR and an even more limited number of patients with severe IR such that these results cannot be considered conclusive; the studies in fact, registrars did not include patients with severe IR or on dialysis. Only some case reports of patients with severe renal insufficiency treated are described in the literature with inhibitory immunocheckpoints without this leading to aggravation of renal function baseline or changes efficacy or toxicity; however few of these reported cases involve patients with metastatic renal cell carcinoma. And' instead, a case of a patient with renal neoplasm in hemodialysis treatment with benefit in terms of objective response from nivolumab therapy. it is also known from the analysis conducted on patients treated with nivolumab within the EAP in Italy, that this drug has a benefit in terms of effectiveness and safety even for older patients, who represent only a small share of the population of pivotal studies; such patients may more frequently have both by age and by comorbidity a reduction in basic renal function. Aim of our retrospective study is to assess whether there are differences in the profile of toxicity in renal cell carcinoma patients treated with Nivolumab in line II or III based on renal function. Patients will be stratified in 3 patient groups:

* patients with normal or mildly reduced renal function (GFR<90 and ≥60 ml/min/1.73 m^2);
* patients with moderate renal failure (GFR <60 e ≥30 ml/min/1.73 m^2),
* patients with severe renal failure (GFR <30 e ≥15 ml/min/1.73 m^2).

ELIGIBILITY:
Inclusion Criteria:

* signing informed consent, in case of patients still alive;
* histologically confirmed diagnosis of metastatic renal cell carcinoma;
* at least one administration of Nivolumab therapy, in the second-or third line of treatment february 2017 to December 31, 2018;
* availability of inpatient and/or outpatient medical records for clinical data collection.

Exclusion Criteria:

* patients who have received immunotherapy under EAP (Expanded Access Programm) or other clinical trials;
* dialysis patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affered to the structures involved treated with at least one administration of the drug Nivolumab line II or III for metastatic renal cell carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events | At study completion (up to 16 months)
  To describe the safety of the treatment, the number of adverse events will be counted percentage, grade 1-2 and 3-4 and will compare for the 3 patient stratification groups.

SECONDARY OUTCOMES:
Effectiveness of the treatment | At study completion (up to 16 months)
  The effectiveness of treatment in the population in terms of objective responses will be described (ORR) defined as number of patients in complete response, partial response established by clinicians according to RECIST 1.1 criteria. Objective response rates will be compared between the three groups of patient stratification.
Survival assessment | At study completion (up to 16 months)
  It will describe the possible correlation between the three patient stratification groups and the survival. The overall survival estimate is defined as the time from treatment start date to date of death from any cause. Survival time comes discontinued at the date of the last follow-up visit for patients alive or lost to follow-up.
Evaluation of progression free time | At study completion (up to 16 months)
  The possible correlation between the three patient stratification groups and the progression free survival (PFS) will be described. The PFS estimate is defined as the time from the start date of treatment at the date of disease progression. Time to progression is interrupted at date of last follow-up visit for patients not progressed.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Italy

REFERENCES:
- [Background] Masini C, Vitale MG, Maruzzo M, Procopio G, de Giorgi U, Buti S, Rossetti S, Iacovelli R, Atzori F, Cosmai L, Vignani F, Prati G, Scagliarini S, Guida A, Berselli A, Pinto C. Safety and Efficacy of Pazopanib in First-Line Metastatic Renal-Cell Carcinoma With or Without Renal Failure: CORE-URO-01 Study. Clin Genitourin Cancer. 2019 Feb;17(1):e150-e155. doi: 10.1016/j.clgc.2018.10.001. Epub 2018 Oct 10. PMID 30396828
- [Background] Gupta S, Parsa V, Heilbrun LK, Smith DW, Dickow B, Heath E, Vaishampayan U. Safety and efficacy of molecularly targeted agents in patients with metastatic kidney cancer with renal dysfunction. Anticancer Drugs. 2011 Sep;22(8):794-800. doi: 10.1097/CAD.0b013e328346af0d. PMID 21799472
- [Background] Wanchoo R, Karam S, Uppal NN, Barta VS, Deray G, Devoe C, Launay-Vacher V, Jhaveri KD; Cancer and Kidney International Network Workgroup on Immune Checkpoint Inhibitors. Adverse Renal Effects of Immune Checkpoint Inhibitors: A Narrative Review. Am J Nephrol. 2017;45(2):160-169. doi: 10.1159/000455014. Epub 2017 Jan 12. PMID 28076863
- [Background] Vitale MG, Scagliarini S, Galli L, Pignata S, Lo Re G, Berruti A, Defferrari C, Spada M, Masini C, Santini D, Ciuffreda L, Ruggeri EM, Bengala C, Livi L, Fagnani D, Bonetti A, Giustini L, Hamzaj A, Procopio G, Caserta C, Sabbatini R. Efficacy and safety data in elderly patients with metastatic renal cell carcinoma included in the nivolumab Expanded Access Program (EAP) in Italy. PLoS One. 2018 Jul 6;13(7):e0199642. doi: 10.1371/journal.pone.0199642. eCollection 2018. PMID 29979712
- [Background] Carlo MI, Feldman DR. Response to Nivolumab in a Patient With Metastatic Clear Cell Renal Cell Carcinoma and End-stage Renal Disease on Dialysis. Eur Urol. 2016 Dec;70(6):1082-1083. doi: 10.1016/j.eururo.2016.05.040. Epub 2016 Jun 13. No abstract available. PMID 27311362
- [Background] Herz S, Hofer T, Papapanagiotou M, Leyh JC, Meyenburg S, Schadendorf D, Ugurel S, Roesch A, Livingstone E, Schilling B, Franklin C. Checkpoint inhibitors in chronic kidney failure and an organ transplant recipient. Eur J Cancer. 2016 Nov;67:66-72. doi: 10.1016/j.ejca.2016.07.026. Epub 2016 Sep 8. PMID 27614165
- [Background] Motzer RJ, Tannir NM, McDermott DF, Aren Frontera O, Melichar B, Choueiri TK, Plimack ER, Barthelemy P, Porta C, George S, Powles T, Donskov F, Neiman V, Kollmannsberger CK, Salman P, Gurney H, Hawkins R, Ravaud A, Grimm MO, Bracarda S, Barrios CH, Tomita Y, Castellano D, Rini BI, Chen AC, Mekan S, McHenry MB, Wind-Rotolo M, Doan J, Sharma P, Hammers HJ, Escudier B; CheckMate 214 Investigators. Nivolumab plus Ipilimumab versus Sunitinib in Advanced Renal-Cell Carcinoma. N Engl J Med. 2018 Apr 5;378(14):1277-1290. doi: 10.1056/NEJMoa1712126. Epub 2018 Mar 21. PMID 29562145
- [Background] Motzer RJ, Escudier B, McDermott DF, George S, Hammers HJ, Srinivas S, Tykodi SS, Sosman JA, Procopio G, Plimack ER, Castellano D, Choueiri TK, Gurney H, Donskov F, Bono P, Wagstaff J, Gauler TC, Ueda T, Tomita Y, Schutz FA, Kollmannsberger C, Larkin J, Ravaud A, Simon JS, Xu LA, Waxman IM, Sharma P; CheckMate 025 Investigators. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13. doi: 10.1056/NEJMoa1510665. Epub 2015 Sep 25. PMID 26406148
- [Background] Choueiri TK, Escudier B, Powles T, Mainwaring PN, Rini BI, Donskov F, Hammers H, Hutson TE, Lee JL, Peltola K, Roth BJ, Bjarnason GA, Geczi L, Keam B, Maroto P, Heng DY, Schmidinger M, Kantoff PW, Borgman-Hagey A, Hessel C, Scheffold C, Schwab GM, Tannir NM, Motzer RJ; METEOR Investigators. Cabozantinib versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1814-23. doi: 10.1056/NEJMoa1510016. Epub 2015 Sep 25. PMID 26406150
- [Background] Decastro GJ, McKiernan JM. Epidemiology, clinical staging, and presentation of renal cell carcinoma. Urol Clin North Am. 2008 Nov;35(4):581-92; vi. doi: 10.1016/j.ucl.2008.07.005. PMID 18992612
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998